CLINICAL TRIAL: NCT04041115
Title: Effect of a Multifactorial Intervention (Non-alcoholic Beer, Diet and Exercise) on Endothelial Function, Nutritional Status and Quality of Life in Patients With Cirrhosis
Brief Title: Effect of Non-alcoholic Beer in Cirrhosis
Acronym: LFN-NAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICTLAN-2
Record Dates: First submitted 2019-04-26; First posted 2019-08-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2019-03

CONDITIONS: Endothelial Dysfunction; Nutritional Status; Quality of Life
Keywords: cirrhosis; nutrition; sarcopenia; non-alcoholic beer
MeSH Terms: conditions — Fibrosis; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): personalized nutritional therapy + aerobic exercise
  Interventions: Other: control
- Non-alcoholic Beer (Active Comparator): non-alcoholic beer + personalized nutritional therapy + aerobic exercise
  Interventions: Dietary Supplement: Non-alcoholic beer

INTERVENTIONS:
Dietary Supplement: Non-alcoholic beer — Treatment consisted of 330ml non-alcoholic beer per day, plus an individualized dietary program and an exercise program with a pedometer-based bracelet to reach at least 5000 steps/day during 2 + 8 weeks.
  Arms: Non-alcoholic Beer
Other: control — Treatment consisted of 330ml of water, plus an individualized dietary program and an exercise program with a pedometer-based bracelet to reach at least 5000 steps/day during 2 + 8 weeks.
  Arms: Control

SUMMARY:
The implementation of nutritional strategies targeting several variables at once could benefit patients with cirrhosis. Non-alcoholic beer has different compounds derived from hops that exert antioxidant, anti-inflammatory and nutritional properties. The aim of this study is to evaluate the effect of diet + exercise and non-alcoholic beer on nutritional status, endothelial function and quality of life in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Liver Cirrhosis of any aetiology (liver biopsy or a combination of clinical and biochemical variables plus evidence of portal hypertension); without decompensation during the past month; serum creatinine <1.5 mg%; able to attend the appointed visits and willing to participate in the study.

Exclusion Criteria:

* Severe concomitant cardiopulmonary diseases; decompensated type 2 Diabetes Mellitus, insulin use or proliferative diabetic retinopathy; orthopedic or osteomuscular limitations; any type of cancer; primary sclerosing cholangitis and inflammatory bowel disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 8 weeks
  improvement in impedance-derived phase angle (PhA)
Endothelial function | 8 weeks
  improvement in flow-mediated dilation (brachial artery)
Endothelial dysfunction | 8 weeks
  improvement in serum markers of endothelial function (v.gr. nitric oxide, NO; prostacyclin, PGI2, etc.)
Quality of life questionnaire | 8 weeks
  Improvement in quality of life questionnaire CLDQ (chronic liver disease questionnaire)
Changes in the heterogeneity of gut Microbiota | 8 weeks
  Changes in the heterogeneity of fecal microbiota in terms of bacterial diversity will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo U. Macías-Rodríguez, M.D., Ph.D., Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran